CLINICAL TRIAL: NCT03662451
Title: Single Site Versus Multi Site Robotic Hysterectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Hospital never started on single site laparoscopy
Sponsor: Herning Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Finn Lauszus, Associate professor, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Single site robot study
Record Dates: First submitted 2018-06-07; First posted 2018-09-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Rehabilitation; Pain, Postoperative; Wound Infection
Keywords: Return-to-work; Cosmesis; Visual analogue pain score
MeSH Terms: conditions — Pain, Postoperative; Wound Infection

STUDY DESIGN:
Intervention Model Description: Women are randomized to either robotic single site or multi site hysterectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic single-site hysterectomy (Active Comparator): Robotic single-site hysterectomy is performed in this arm
  Interventions: Procedure: Robotic assisted hysterectomy
- Robotic multi-site hysterectomy (Active Comparator): Robotic multi-site hysterectomy is performed in this arm
  Interventions: Procedure: Robotic assisted hysterectomy

INTERVENTIONS:
Procedure: Robotic assisted hysterectomy — Periumbilical single incision vs multiple abdominal incisions for hysterectomy

SUMMARY:
Robotic single site surgery (R-SSH) is a novel technique, which may be superior to multi site hysterectomy (R-MSH) in select patients regarding cosmesis and postoperative pain. A randomized trial is performed to compare R-SSH with R-MSH with regard to the postoperative rehabilitation, cosmesis, the operational cost, and the perioperative morbidity.

DETAILED DESCRIPTION:
The study is scheduled to start November 2018 and compares robotic single site to multi site hysterectomy. Procedures are performed on two locations, Herning and Herlev Hospitals, by experienced surgeons. Patients are randomized to either R-SSH (No.=62) or R-MSH (No.=62). Patient's satisfaction with body image and cosmesis is assessed at different time points pre- and postoperatively by means of validated cosmesis scales and Body Image Questionnaire and photo-evaluations.

Postoperative pain and split times spent at the operation theatre will be registered as secondary outcome parameters.

A follow-up at 1, 3 and 6 month include evaluation of the scar and registration of port-site hernias and vaginal dehiscence or other complications. Interviews and diaries will include time of return to home and work, daily activities including sexuality The R-SSH is performed using da Vinci, Xi robotic system. One single port, diameter 2 cm is applied. Applying an additional assistant port is defined conversion of procedure R-MSH is performed using standard equipment and 4 trocars, 5 mm each.

Sample size calculation was based a previous study on fast track hysterectomy, which showed a difference in return to work of 4 days. 62 women in each group is needed with standard deviation ±8 and a power of 80%. To include those not working, the calculation was performed with an expected visual analog pain score of 0.86 ±0.2 and 62 in each group and suggested that the sample was sufficient to detect of difference of 0.1 in visual analog pain score with a power of 80%. All calculation are based on two-sided testing with alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy on benign indication,
* American Society of Anesthetists group 1 or 2,
* BMI less than 30 kg/m2
* uterine size less than 300 g estimated by ultrasound, using Ferraris formula.

Exclusion Criteria:

* adhesions
* prior extensive abdominal surgery
* prior midline incision
* cutis laxa of abdomen surgery
* endometriosis
* more than 1 cesarean section
* malignant disease

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-10-16 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Scar appearance and satisfaction | Six months after operation
  Appearance and evaluation of scar by POSAS scale (see www.posas.org and reference below) which has a scale from 1-10, where 1 is minimum and 10 is maximum; on scar's pain, its itching, on difference from normal skin, on stiffness, on thickness, on irregularity and general satisfaction

SECONDARY OUTCOMES:
Scoring of abdominal pain | Visual analogue pain score at first, second, third, fourth, fifth, and sixth month after operation
  Visual analogue pain score with a minimum '0' and maximum '10'

CONTACTS AND LOCATIONS:
Overall Officials: Finn F Lauszus, PhD, Principal Investigator — Herning Hospital
Locations (1):
- Gynecology Dept. Herning Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Awaiting consensus in the steering Group on meeting, posters, abstracts, and publications

REFERENCES:
- [Background] El Hachem L, Andikyan V, Mathews S, Friedman K, Poeran J, Shieh K, Geoghegan M, Gretz HF 3rd. Robotic Single-Site and Conventional Laparoscopic Surgery in Gynecology: Clinical Outcomes and Cost Analysis of a Matched Case-Control Study. J Minim Invasive Gynecol. 2016 Jul-Aug;23(5):760-8. doi: 10.1016/j.jmig.2016.03.005. Epub 2016 Mar 15. PMID 26992935
- [Background] Golkar FC, Ross SB, Sperry S, Vice M, Luberice K, Donn N, Morton C, Hernandez JM, Rosemurgy AS. Patients' perceptions of laparoendoscopic single-site surgery: the cosmetic effect. Am J Surg. 2012 Nov;204(5):751-61. doi: 10.1016/j.amjsurg.2011.07.026. PMID 23140831
- [Background] Sandberg EM, la Chapelle CF, van den Tweel MM, Schoones JW, Jansen FW. Laparoendoscopic single-site surgery versus conventional laparoscopy for hysterectomy: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 May;295(5):1089-1103. doi: 10.1007/s00404-017-4323-y. Epub 2017 Mar 29. PMID 28357561
- [Background] Yeung PP Jr, Bolden CR, Westreich D, Sobolewski C. Patient preferences of cosmesis for abdominal incisions in gynecologic surgery. J Minim Invasive Gynecol. 2013 Jan-Feb;20(1):79-84. doi: 10.1016/j.jmig.2012.09.008. PMID 23312246
- [Background] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233